CLINICAL TRIAL: NCT04796779
Title: The Pediatric Artificial Pancreas (PEDAP) Trial: A Randomized Controlled Comparison of the Control-IQ Technology Versus Standard of Care in Young Children in Type 1 Diabetes
Brief Title: The Pediatric Artificial Pancreas (PEDAP) Trial of Control-IQ Technology in Young Children in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Breton (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Marc Breton, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200433; 1U01DK127551-01 (NIH); RFA-DK-19-036 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2021-02-15; First posted 2021-03-15 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Type 1 Diabetes
Keywords: Control-IQ Technology; Insulin Pump; Closed Loop Control (CLC); Continuous Glucose Monitor (CGM); Multiple Daily Injections (MDI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CLC Group (Experimental): Participants who skip or successfully complete the run-in will be randomly assigned 2:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs Standard of Care (SC group) for 3 weeks. Participants randomized to the intervention group will use the Tandem t:slim X2 with Control-IQ Technology v1.0 during the first 13 weeks of the study (RCT phase, weeks 1-13) and then use Tandem t:slim X2 insulin pump with Control-IQ Technology v1.5 for the remaining 13 weeks of the study (extension phase, weeks 14-26).
  Interventions: Device: Tandem t:slim X2 with Control-IQ Technology Pro; Device: Tandem t:slim X2 with Control-IQ Technology V1.5
- SC Group (Active Comparator): Participants who skip or successfully complete the run-in will be randomly assigned 2:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs Standard of Care (SC group) for 3 weeks. Participants randomized to the SC group will use their existing insulin therapy in conjunction with study Dexcom G6 CGM during the first 13 weeks of the study (RCT phase, weeks 1-13). The SC group will then transition to using the Tandem t:slim X2 insulin pump with Control-IQ Technology v1.5 and study Dexcom G6 CGM for the remaining 13 weeks of the study (weeks 14-26).
  Interventions: Device: Standard Care (SC); Device: Tandem t:slim X2 with Control-IQ Technology V1.5

INTERVENTIONS:
Device: Tandem t:slim X2 with Control-IQ Technology Pro — The Tandem t:slim X2 with Control-IQ Technology Pro is an "artificial pancreas" (AP) application that uses advanced closed loop control algorithms to automatically manage blood glucose levels for people with Type 1 Diabetes. The system modulates insulin to keep blood glucose in a targeted range. The system components include the t:slim X2 with Control-IQ Technology and the Dexcom G6 CGM. The system is very similar to the commercially available t:sli X2 with Control-IQ but modified to accept the lower weight and Total Daily Insulin of the studied population.
  Arms: CLC Group
Device: Standard Care (SC) — Standard of Care consists in the participant existing insulin therapy (prior to enrollment) in conjunction with a study Dexcom G6 CGM. Existing insulin therapies are defined as multiple daily injections of insulin (MDI) or use of an insulin pump without hybrid closed-loop control capabilities (low-glucose suspend or predictive low-glucose suspend functionality is permitted).
  Arms: SC Group
Device: Tandem t:slim X2 with Control-IQ Technology V1.5 — The Tandem t:slim X2 with Control-IQ Technology V1.5 is an "artificial pancreas" (AP) application that uses advanced closed loop control algorithms to automatically manage blood glucose levels for people with Type 1 Diabetes. The system modulates insulin to keep blood glucose in a targeted range. The system components include the t:slim X2 with Control-IQ Technology and the Dexcom G6 CGM. The system is derived from the commercially available t:slim X2 with Control-IQ, with additional features.

SUMMARY:
The purpose of this study is to learn whether an investigational automated insulin delivery system ("study system") for young children (2 yo to less than 6 yo) with type 1 diabetes can safely improve blood glucose (sometimes called blood sugar) control.

DETAILED DESCRIPTION:
Participants will be randomized to closed loop control (CLC) system (t:slim X2 with Control-IQ Technology) or to standard of care where the children will continue to use his or her personal insulin pump or multiple daily injections. Both groups will use a continuous glucose monitor (CGM) throughout the study. The study system will also use a study insulin pump and a software algorithm to automatically give insulin and control blood glucose. This system is also sometimes called a "closed-loop" system.

This study will take about 6-7 months for the child to complete. Study visits can be completed from home via videoconference (e.g. Zoom) without visiting the clinic or in-person at the clinic.

A subset of participants will be asked to join an ancillary study with Meal Bolus and Exercise challenges during the extension phase. Data collected from the start of each of these challenges until the following morning will be excluded from the analysis of the extension phase.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least 6 months and using insulin for at least 6 months
2. Familiarity and use of a carbohydrate ratio for meal boluses.
3. Age ≥2 and <6 years old
4. Living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff.
5. Investigator has confidence that the parent can successfully operate all study devices and is capable of adhering to the protocol
6. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study for participants using a study-provided Tandem pump during the study.

   • Study will not be providing insulin; therefore, participants will need to have access to either lispro or aspart
7. Total daily insulin dose (TDD) at least 5 U/day
8. Body weight at least 20 lbs.
9. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (see section 2.3)
10. Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff.
11. Parent/guardian proficient in reading and writing English.

Exclusion Criteria:

1. Concurrent use of any non-insulin glucose-lowering agent (including Glucagon-like peptide-1 [GLP-1] agonists, Symlin, Dipeptidyl peptidase-4 [DPP-4] inhibitors, Sodium-glucose Cotransporter-2 (SGLT-2) inhibitors, sulfonylureas).
2. Hemophilia or any other bleeding disorder
3. History of >1 severe hypoglycemic event with seizure or loss of consciousness in the last 3 months
4. History of >1 DKA event in the last 6 months not related to illness, infusion set failure, or initial diagnosis
5. History of chronic renal disease or currently on hemodialysis
6. History of adrenal insufficiency
7. Hypothyroidism that is not adequately treated
8. Use of oral or injectable steroids within the last 8 weeks
9. Known, ongoing adhesive intolerance
10. Plans to receive blood transfusions or erythropoietin injections during the course of the study
11. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk (specified in the study procedure manual)
12. Currently using any closed-loop system, or using an insulin pump that is incompatible with use of the study CGM
13. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
14. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lum, MS, Study Director — Jaeb Center for Health Research
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available after the primary publications of each study.

REFERENCES:
- [Background] Wadwa RP, Reed ZW, Buckingham BA, DeBoer MD, Ekhlaspour L, Forlenza GP, Schoelwer M, Lum J, Kollman C, Beck RW, Breton MD; PEDAP Trial Study Group. Trial of Hybrid Closed-Loop Control in Young Children with Type 1 Diabetes. N Engl J Med. 2023 Mar 16;388(11):991-1001. doi: 10.1056/NEJMoa2210834. PMID 36920756
- [Derived] Beck RW, Kanapka LG, Breton MD, Brown SA, Wadwa RP, Buckingham BA, Kollman C, Kovatchev B. A Meta-Analysis of Randomized Trial Outcomes for the t:slim X2 Insulin Pump with Control-IQ Technology in Youth and Adults from Age 2 to 72. Diabetes Technol Ther. 2023 May;25(5):329-342. doi: 10.1089/dia.2022.0558. Epub 2023 Apr 12. PMID 37067353
- See also: Study Results — https://pubmed.ncbi.nlm.nih.gov/36920756/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CLC Group | SC Group
Started | 68 | 34
Completed | 67 | 34
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLC Group | SC Group | Total
Number analyzed (Participants) | 68 | 34 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.84 (1.23) | 4.06 (1.25) | 3.92 (1.24)
Age, Customized [Count of Participants; unit: Participants]
  2 to <4 years | 31 | 16 | 47
  4 to <6 years | 37 | 18 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 19 | 52
  Male | 35 | 15 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 50 | 25 | 75
  Black/African American | 4 | 2 | 6
  Hispanic or Latino | 11 | 5 | 16
  Asian | 1 | 1 | 2
  More than one race | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 68 | 34 | 102
Diabetes Duration [Count of Participants; unit: Participants]
  0.5 to <1 years | 29 | 10 | 39
  1 to <2 years | 24 | 15 | 39
  2 to <4 years | 11 | 7 | 18
  ≥4 years | 4 | 2 | 6
Glycosylated Hemoglobin (HbA1c) at Randomization [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — Population: Missing data (CLC/SC): HbA1c 4/2
  Percentage of glycosylated hemoglobin
    number analyzed (Participants) | 64 | 32 | 96
    (all) | 7.5 (1.2) | 7.7 (0.9) | 7.6 (1.1)
Insulin Modality [Count of Participants; unit: Participants]
  Insulin pump | 42 | 24 | 66
  Multiple daily injections | 26 | 10 | 36
Prior Continuous Glucose Monitor (CGM) Use [Count of Participants; unit: Participants]
  In past, but not current | 2 | 0 | 2
  Current | 66 | 34 | 100
Annual Household Income [Count of Participants; unit: Participants] — Population: Missing data (CLC/SC): annual household income 4/2
  Participants
    number analyzed (Participants) | 64 | 32 | 96
    $25,000 - <$35,000 | 2 | 2 | 4
    $35,000 - <$50,000 | 6 | 4 | 10
    $50,000 - <$75,000 | 8 | 5 | 13
    $75,000 - <$100,000 | 11 | 7 | 18
    $100,000 - <$200,000 | 22 | 10 | 32
    ≥ $200,000 | 15 | 4 | 19
Parent Education [Count of Participants; unit: Participants]
  ≤High School Diploma | 6 | 3 | 9
  Associates Degree or Some College but no Degree | 2 | 1 | 3
  Bachelor's Degree | 6 | 5 | 11
  Master's Degree | 22 | 13 | 35
  Doctoral or Prof Degree | 32 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Time in Range
Description: Time in range is the amount of time spent in the target glucose range-between 70 and 180 mg/dL-as measured by CGM
Time Frame: 13 weeks
Population: One participant in the CLC group was missing baseline CGM data.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | CLC Group | SC Group
Number analyzed (Participants) | 68 | 34
Percent of time
  Baseline: number analyzed (Participants) | 67 | 34
  Baseline | 56.7 (18.0) | 54.9 (14.7)
  Week 13 | 69.3 (11.1) | 55.9 (12.6)
Statistical Analysis 1: Comparison: CLC Group vs SC Group; Test type: Superiority; p < 0.001, Direct likelihood model; The model was adjusted for the baseline value of the metric, age, prior CGM and pump use, and site as a random effect

2. Secondary Outcome: CGM-measured Percent Above 250 mg/dL
Description: Percentage of time with a glucose above 250 mg/dL as measured by CGM
Time Frame: 13 weeks
Population: One participant in the CLC group was missing baseline CGM data.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | CLC Group | SC Group
Number analyzed (Participants) | 68 | 34
Percent of time
  Baseline: number analyzed (Participants) | 67 | 34
  Baseline | 14.8 (15.5) | 16.0 (13.9)
  Week 13 | 8.4 (7.2) | 15.0 (10.9)
Statistical Analysis 1: Comparison: CLC Group vs SC Group; Test type: Superiority; p < 0.001, Robust regression using M-estimation — To preserve the overall type I error for the multiple secondary outcomes, a hierarchical gatekeeping approach was used; The model was adjusted for baseline value of the metric, age, prior CGM and pump use, and site as a fixed effect

3. Secondary Outcome: CGM-measured Mean Glucose
Description: Average glucose value measured by CGM
Time Frame: 13 weeks
Population: One participant in the CLC group was missing baseline CGM data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CLC Group | SC Group
Number analyzed (Participants) | 68 | 34
mg/dL
  Baseline: number analyzed (Participants) | 67 | 34
  Baseline | 173 (36) | 176 (26)
  Week 13 | 155 (20) | 174 (22)
Statistical Analysis 1: Comparison: CLC Group vs SC Group; Test type: Superiority; p < 0.001, Direct likelihood model — To preserve the overall type I error for the multiple secondary outcomes, a hierarchical gatekeeping approach was used; The model was adjusted for the baseline value of the metric, age, prior CGM and pump use, and site as a random effect

4. Secondary Outcome: HbA1c at 13 Weeks
Description: HbA1c at 13 weeks
Time Frame: 13 weeks
Population: Baseline HbA1c values were available for n=64/68 in the CLC group and n=32/34 in the SC group. At 13 Weeks, HbA1c data were available for n=62/68 in the CLC group and n=33/34 in the SC group.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | CLC Group | SC Group
Number analyzed (Participants) | 68 | 34
Percentage of glycosylated hemoglobin
  Baseline: number analyzed (Participants) | 64 | 32
  Baseline | 7.5 (1.2) | 7.7 (0.9)
  Week 13: number analyzed (Participants) | 62 | 33
  Week 13 | 7.0 (0.8) | 7.5 (0.9)
Statistical Analysis 1: Comparison: CLC Group vs SC Group; Test type: Superiority; p < 0.001, Direct likelihood model — To preserve the overall type I error for the multiple secondary outcomes, a hierarchical gatekeeping approach was used; The model was adjusted for the baseline value of the metric, age, prior CGM and pump use, and site as a random effect

5. Secondary Outcome: CGM-measured Percent Below 70 mg/dL
Description: Percentage of time with glucose below 70 mg/dL as measured by CGM
Time Frame: 13 weeks
Population: One participant in the CLC group was missing baseline CGM data.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | CLC Group | SC Group
Number analyzed (Participants) | 68 | 34
Percent of time
  Baseline: number analyzed (Participants) | 67 | 34
  Baseline | 3.0 (2.2) | 2.7 (2.0)
  Week 13 | 3.0 (1.8) | 3.0 (2.2)
Statistical Analysis 1: Comparison: CLC Group vs SC Group; Test type: Superiority; p = 0.57, Robust regression using M-estimation — To preserve the overall type I error for the multiple secondary outcomes, a hierarchical gatekeeping approach was used; The model was adjusted for the baseline value of the metric, age, prior CGM and pump use, and site as a fixed effect

6. Secondary Outcome: CGM-measured Percent Below 54 mg/dL
Description: Percentage of time with glucose below 54 mg/dL as measured by CGM
Time Frame: 13 weeks
Population: One participant in the CLC group was missing baseline CGM data.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | CLC Group | SC Group
Number analyzed (Participants) | 68 | 34
Percent of time
  Baseline: number analyzed (Participants) | 67 | 34
  Baseline | 0.6 (0.7) | 0.5 (0.6)
  Week 13 | 0.6 (0.5) | 0.5 (0.5)

7. Other Pre Specified Outcome: Percent Above 180 mg/dL
Description: percent above 180 mg/dL
Time Frame: 13 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percent in Range 70-140 mg/dL
Description: percent in range 70-140 mg/dL
Time Frame: 13 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Glucose Variability Measured With the Coefficient of Variation (CV)
Description: glucose variability measured with the coefficient of variation (CV)
Time Frame: 13 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Glucose Variability Measured With the Standard Deviation (SD)
Description: glucose variability measured with the standard deviation (SD)
Time Frame: 13 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: CGM-measured Percent <60 mg/dL
Description: CGM-measured percent <60 mg/dL
Time Frame: 13 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Low Blood Glucose Index (LBGI)*
Description: low blood glucose index (LBGI)*
Time Frame: 13 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Hypoglycemic Events (Defined as at Least 15 Consecutive Minutes <54 mg/dL)
Description: hypoglycemic events (defined as at least 15 consecutive minutes <54 mg/dL)
Time Frame: 13 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Hyperglycemic Events (Defined as at Least 90 Consecutive Minutes >300 mg/dL)
Description: hyperglycemic events (defined as at least 90 consecutive minutes >300 mg/dL)
Time Frame: 13 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Percent >300 mg/dL
Description: percent >300 mg/dL
Time Frame: 13 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: High Blood Glucose Index (HBGI)*
Description: high blood glucose index (HBGI)*
Time Frame: 13 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Percent in Range 70-180 mg/dL Improvement From Baseline to 13 Weeks ≥5 Percent
Description: percent in range 70-180 mg/dL improvement from baseline to 13 weeks ≥5 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Percent in Range 70-180 mg/dL Improvement From Baseline to 13 Weeks ≥10 Percent
Description: percent in range 70-180 mg/dL improvement from baseline to 13 weeks ≥10 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Percent Time in Range 70-180 mg/dL >70 Percent and Percent Time <70 mg/dL <4 Percent
Description: percent time in range 70-180 mg/dL >70 percent and percent time <70 mg/dL <4 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: HbA1c <7.0 Percent at 13 Weeks
Description: HbA1c <7.0 percent at 13 weeks
Time Frame: 13 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: HbA1c <7.5 Percent at 13 Weeks
Description: HbA1c <7.5 percent at 13 weeks
Time Frame: 13 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: HbA1c Improvement From Baseline to 13 Weeks >0.5 Percent
Description: HbA1c improvement from baseline to 13 weeks >0.5 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: HbA1c Improvement From Baseline to 13 Weeks >1.0 Percent
Description: HbA1c improvement from baseline to 13 weeks >1.0 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

24. Other Pre Specified Outcome: HbA1c Relative Improvement From Baseline to 13 Weeks >10 Percent
Description: HbA1c relative improvement from baseline to 13 weeks >10 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

25. Other Pre Specified Outcome: HbA1c Absolute Improvement From Baseline to 13 Weeks >1.0 Percent or HbA1c <7.0 Percent at 13 Weeks
Description: HbA1c absolute improvement from baseline to 13 weeks >1.0 percent or HbA1c <7.0 percent at 13 weeks
Time Frame: 13 weeks
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Number of Severe Hypoglycemic (SH) Events and SH Event Rate Per 100 Person-years
Description: Number of SH events and SH event rate per 100 person-years
Time Frame: 13 weeks
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Number of Diabetic Ketoacidosis (DKA) Events and DKA Event Rate Per 100 Person-years
Description: Number of DKA events and DKA event rate per 100 person-years
Time Frame: 13 weeks
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Number of Other Serious Adverse Events
Description: Number of other serious adverse events (SAEs other than SH events and DKA events)
Time Frame: 13 weeks
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Any Adverse Event Rate
Description: Any adverse event rate
Time Frame: 13 weeks
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Number of Calendar Days With Any Ketone Level ≥1.0 mmol/L (if ≥5 Total Calendar Days Combined)
Description: Number of calendar days with any ketone level ≥1.0 mmol/L (if ≥5 total calendar days combined)
Time Frame: 13 weeks
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Worsening of HbA1c From Baseline to 13 Weeks by >0.5 Percent
Description: Worsening of HbA1c from baseline to 13 weeks by >0.5 percent
Time Frame: 13 weeks
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Adverse Device Effects (ADE)
Description: Adverse device effects (ADE) in intervention group only
Time Frame: 13 weeks
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Serious Adverse Device Events (SADE)
Description: Serious adverse device events (SADE) in intervention group only
Time Frame: 13 weeks
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Unanticipated Adverse Device Effects (UADE)
Description: Unanticipated adverse device effects (UADE) in intervention group only
Time Frame: 13 weeks
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Total Daily Insulin (Units/kg)
Description: Total daily insulin (units/kg)
Time Frame: 13 weeks
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Percentage of Total Insulin Delivered Via Basal
Description: Percentage of total insulin delivered via basal
Time Frame: 13 weeks
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Weight
Description: Weight
Time Frame: 13 weeks
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI)
Time Frame: 13 weeks
Reporting Status: Not Posted

39. Other Pre Specified Outcome: PedsQL Diabetes Module - Total Score and 5 Subscales
Description: PedsQL Diabetes Module - total score and 5 subscales: Diabetes, Treatment 1, Treatment 2, Worry, Communication
Time Frame: 13 weeks
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Pediatric Inventory for Parents (PIP) 2 Domains Each With a Total Score and 4 Subscales for (5x2=10 Difference Scores)
Description: Pediatric Inventory for Parents (PIP) 2 domains each with a total score and 4 subscales for (5x2=10 difference scores): Frequency (Total Score, Communication, Medical Care, Role Function, Emotional Functioning), Difficulty ( Same total + 4 subscales as above for frequency)
Time Frame: 13 weeks
Reporting Status: Not Posted

41. Other Pre Specified Outcome: INSPIRE Survey (Insulin Delivery Systems: Perceptions, Ideas, Reflections and Expectations) (CLC Arm Only)
Description: INSPIRE (CLC arm only) 5-point Likert scale from strongly agree to strongly disagree, along with an N/A option.
Time Frame: 13 weeks
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (PSQI) Global Score
Description: An abbreviated 9-question version of the Pittsburgh Sleep Quality Index (PSQI), a validated tool for assessing self-reported sleep quantity and quality, will be completed by parents. Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: 13 weeks
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Fear of Hypoglycemia Survey for Parents (HFS-P) - Total Score, 2 Subscales and 4 Factor Scores
Description: Fear of Hypoglycemia Survey for Parents (HFS-P) - total score, 2 subscales and 4 factor scores: Behavior (avoidance, Maintain high BG), Worry (Helplessness, Social consequences)
Time Frame: 13 weeks
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Number of SH Events During, Immediately After and Overnight From the Study Challenges
Description: Number of SH events during, immediately after and overnight from the study challenges
Time Frame: Up to 24 hour period
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Number of Adverse Events During, Immediately After and Overnight From the Study Challenges
Description: Number of adverse events during, immediately after and overnight from the study challenges
Time Frame: Up to 24 hour period
Reporting Status: Not Posted

46. Other Pre Specified Outcome: CGM-measured % <54 mg/dL Overnight (All Challenge Types)
Description: CGM-measured % <54 mg/dL overnight (all challenge types)
Time Frame: 8 hours
Reporting Status: Not Posted

47. Other Pre Specified Outcome: CGM-measured % <70 mg/dL Overnight (All Challenge Types)
Description: CGM-measured % <70 mg/dL overnight (all challenge types)
Time Frame: 8 hours
Reporting Status: Not Posted

48. Other Pre Specified Outcome: CGM-measured % >180 mg/dL Overnight (All Challenge Types)
Description: CGM-measured % >180 mg/dL overnight (all challenge types)
Time Frame: 8 hours
Reporting Status: Not Posted

49. Other Pre Specified Outcome: CGM-measured % <54 mg/dL During the Two Hours Immediately Following the Start of Exercise for Each Exercise-related Challenge
Description: CGM-measured % <54 mg/dL during the two hours immediately following the start of exercise for each exercise-related challenge
Time Frame: 2 hours
Reporting Status: Not Posted

50. Other Pre Specified Outcome: CGM-measured % <70 mg/dL During the Two Hours Immediately Following the Start of Exercise for Each Exercise-related Challenge
Description: CGM-measured % <70 mg/dL during the two hours immediately following the start of exercise for each exercise-related challenge
Time Frame: 2 hours
Reporting Status: Not Posted

51. Other Pre Specified Outcome: CGM-measured % >180 mg/dL During the Four Hours Following the Announced Meal, or Until the Next Meal Bolus is Given, for the Missed Meal Bolus Challenge
Description: CGM-measured % >180 mg/dL during the four hours following the announced meal, or until the next meal bolus is given, for the missed meal bolus challenge
Time Frame: 4 hours
Reporting Status: Not Posted

52. Other Pre Specified Outcome: CGM-measured % >300 mg/dL During the Four Hours Following the Announced Meal, or Until the Next Meal Bolus is Given, for the Missed Meal Bolus Challenge
Description: CGM-measured % >300 mg/dL during the four hours following the announced meal, or until the next meal bolus is given, for the missed meal bolus challenge
Time Frame: 4 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to Week 13
Arm/Group | CLC Group | SC Group
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/34
Serious Adverse Events (participants affected / at risk) | 3/68 | 2/34
Other Adverse Events (participants affected / at risk) | 40/68 | 9/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLC Group (N=68) | SC Group (N=34)
Severe hypoglycemic event (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other serious adverse event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — One participant in the SC group was hospitalized for an asthma flare
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLC Group (N=68) | SC Group (N=34)
Hyperglycemia with or without Ketosis Related to Study Device (Endocrine disorders) | 26 (39) | 0 (0)
Hyperglycemia with or without Ketosis Not Related to Study Device (Endocrine disorders) | 9 (12) | 7 (8)
Hypoglycemia (not severe) (Endocrine disorders) | 2 (2) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Medical Device Site Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 2 (3) | 0 (0)
Streptococcal Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04796779/Prot_001.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04796779/SAP_003.pdf
  • Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04796779/ICF_004.pdf